CLINICAL TRIAL: NCT03677791
Title: Virtual 360°-Tour in Coronary Computed Tomography - Effects of 360° Virtual Counselling Environment in CCTA Patient's Anxiety and Process Time
Brief Title: Virtual 360°-Tour in Coronary Computed Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KPP12345
Record Dates: First submitted 2018-09-14; First posted 2018-09-19 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Disease; Anxiety; Fear
Keywords: counselling; computed tomography; coronary; CT; virtual; 360; anxiety
MeSH Terms: conditions — Coronary Artery Disease; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: RCT (Randomized controlled trial)
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual 360° intervention (Experimental): counselling in the virtual 360° environment and also counselling in accordance with current practice
  Interventions: Other: Virtual tour in coronary computed tomography - 360° counselling environment
- Control group (Active Comparator): counselling in accordance with current practice
  Interventions: Other: Current practice

INTERVENTIONS:
Other: Virtual tour in coronary computed tomography - 360° counselling environment — Virtual tour in coronary computed tomography - 360° counselling environment for CCTA patients
  Arms: Virtual 360° intervention
Other: Current practice — counselling in accordance with current practice: written patient information letter and verbal counselling at the hospital during the CT-examination
  Arms: Control group

SUMMARY:
The purpose of the study is to evaluate the effectiveness of the virtual 360° counselling environment in the anxiety and process time of the patients coming to CCTA (coronary computed tomography angiography). The virtual, 360° environment 'Virtual 360°-tour in coronary computed tomography' uses 360°- technology based on spherical panorama images and resembles the spaces of the hospital according to the patient's pathway in CT-examination and provides information to the patient at various stages of the pathway.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the effectiveness of the virtual 360° counselling environment in the anxiety and process time of the patients coming to CCTA (coronary computed tomography angiography).

The virtual, 360° environment 'Virtual 360°-tour in coronary computed tomography' uses 360°- technology based on spherical panorama images and resembles the spaces of the hospital according to the patient's pathway in CT-examination and provides information to the patient at various stages of the pathway. Patients who have referred first time to the coronary computed tomography can access the virtual CT examination environment via link before entering the hospital. Using the environment requires a network connection and is possible with a computer, tablet or phone. The environment has digital counselling materials in text, image, animation and video formats in three different virtual spaces/views, the environment and examination are presented via pathway of example 59-year female patient with arterial hypertension and exercise related chest pain (angina pectoris).

ELIGIBILITY:
Inclusion Criteria:

* coming to first coronary computed tomography examination
* adult patient
* able to independently fill in question forms

Exclusion Criteria:

* previous coronary computed tomography
* mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
anxiety measured with State-Trait Anxiety Inventory for adults (STAI) | 1 month
  The STAI meter is a two-part adult anxiety meter developed by Charles D. Spielberger and his research team (1983). It separates situation related anxiety (STATE-A) from character related tendency towards anxiety (TRAIT-A). User evaluates his own current anxiety on a four-step scale with forty questions. The respondents choose from the following options at each question: 1 = no anxiety at all, 2 = slight anxiety, 3 = some anxiety 4 = very much anxiety. Scores range from 20 to 80: mild anxiety 20-39 points, moderate anxiety 40-59 points and strong anxiety 60-80 points.

SECONDARY OUTCOMES:
CCTA Process time | 1 month
  Time between patient enrolled to the CCTA at the hospital and when radiographers marked the cCTA examination ended

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Patients', radiographers' and radiography students' experiences of 360° virtual counselling environment for the coronary computed tomography angiography: A qualitative study — http://doi.org/10.1016/j.radi.2020.09.019